CLINICAL TRIAL: NCT02363348
Title: Efficacy and Safety of L Arginine to Prevent Preeclampsia in High Risk Pregnancies
Brief Title: Efficacy and Safety of L Arginine to Prevent Preeclampsia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Civil Juan I. Menchaca (Other)
Responsible Party: Principal Investigator, Eva Elizabet Camarena Pulido, MD, Hospital Civil Juan I. Menchaca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SSJ1054-11
Record Dates: First submitted 2015-01-27; First posted 2015-02-16 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: Preeclampsia
Keywords: L arginine; Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Arginine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (A) (Placebo Comparator): were administered 5 capsules per day each capsule contained 600 mg of magnesia calcinada. Duration: from week 20th of pregnancy until the end of the same.
  dose was administered as follows: two capsules in the morning at breakfast and three capsules at night in dinner.
  Interventions: Other: Placebo
- L arginine (B) (Experimental): were administered 5 capsules per day each capsule contained 600 mg of L arginine. Duration: from week 20th of pregnancy until the end of the same dose was administered as follows: two capsules in the morning at breakfast and three capsules at night in dinner.
  Interventions: Dietary Supplement: L arginine

INTERVENTIONS:
Dietary Supplement: L arginine — L arginine is a basic amino-acid precursor of nitric oxide main vasodilator.
  Arms: L arginine (B)
Other: Placebo — calcined magnesia
  Arms: Placebo (A)

SUMMARY:
Randomized double-blind controled clinical trial to assess the efficacy and safety of L-arginine to prevent preeclampsia.

applied to pregnant women with risk factors for preeclampsia. the main result was the development of preeclampsia as well as side effects to taking l arginine besides perinatal outcomes

DETAILED DESCRIPTION:
Two groups were formed. one received L arginine 3 grams orally at day from the 20th week of pregnancy. the other group received placebo.

Each three weeks were evaluated in search of high blood pressure and proteinuria.

The follow-up was until the end of pregnancy and two weeks after this

ELIGIBILITY:
Inclusion Criteria:

* one or more risk factors for developing preeclampsia (nulliparous, previous history of preeclampsia, chronic hypertension, BMI ≥30)

Exclusion Criteria:

* pregnant women carriers of chronic renal failure
* pre gestational diabetes
* multiple pregnancy and were removed for some reason they received medication that would interfere with the interpretation of results (aspirin)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2010-08; Primary Completion 2013-08 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
efficacy of L arginine to prevent preeclampsia | from time of randomization until the date of diagnostic of preeclampsia or two weeks after delivery wichever came first. approximalety 20 weeks.
  number of patients with diagnosis of preeclampsia. the diagnostic was performed when they presented arterial blood pressure above 140/90 mm / Hg in the span of 6 hours and accompanied by proteinuria (>300 milligrams in one sample) number of patients with high blood pression and proteinuria (ACOG criteria) The evaluations were performed every three weeks until week 31, then every two weeks until week 35 and weekly until pregnancy ended

SECONDARY OUTCOMES:
perinatal outcome | from time to delivery until two weeks after, approximalety 18 weeks
  number of patients with adverse perinatal outcome: APGAR scale < 7 at five minutes, low weight for gestational age (< 10 percentile) and CAPURRO scale < 37 weeks also the need to enter the neonatal intensive care unit
safety of L arginine | from time of randomization until birth approximalety 18 weeks
  number of patients with adverse reactions and/or any alteration of blood test. participants are awarded a diary which recorded the symptoms that caused them any discomfort. If the discomfort was important it was reported via telephone with the treating physician. the paper was reviewed at each appointment. Blood tests such as blood count, liver function tests and kidney were performed every three weeks in search of alterations in the parameters considered normal by those tests (ACOG criteria)

CONTACTS AND LOCATIONS:
Overall Officials: Guadalupe Panduro, Ph, Study Chair — Hospital Civil Juan I. Menchaca
Locations (1):
- Panduro Baron J Guadalupe, Guadalajara, Jalisco, Mexico

REFERENCES:
- [Background] Johal T, Lees CC, Everett TR, Wilkinson IB. The nitric oxide pathway and possible therapeutic options in pre-eclampsia. Br J Clin Pharmacol. 2014 Aug;78(2):244-57. doi: 10.1111/bcp.12301. PMID 24313856
- [Result] Vadillo-Ortega F, Perichart-Perera O, Espino S, Avila-Vergara MA, Ibarra I, Ahued R, Godines M, Parry S, Macones G, Strauss JF. Effect of supplementation during pregnancy with L-arginine and antioxidant vitamins in medical food on pre-eclampsia in high risk population: randomised controlled trial. BMJ. 2011 May 19;342:d2901. doi: 10.1136/bmj.d2901. PMID 21596735